CLINICAL TRIAL: NCT00364377
Title: The Role of Incretins in the Pathogenesis of Fasting and Postprandial Glucose Metabolism in People With Impaired Fasting Glucose
Brief Title: Incretins in Impaired Fasting Glucose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian Vella, Professor of medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-002673
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-11

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Active Comparator): People with impaired fasting glucose randomized to treatment with sitagliptin 100 mg once daily.
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): People with impaired fasting glucose randomized to treatment with placebo once daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100 mg once daily
  Other Names: Januvia
  Arms: Sitagliptin
Other: Placebo — once daily for duration of the study
  Arms: Placebo

SUMMARY:
People with high fasting glucose can develop type 2 diabetes with the passage of time. This study is being done to determine the effect of a novel medication in people with this elevated fasting glucose. Sitagliptin is a substance that raises levels of a hormone normally found in the blood. This hormone, called glucagon-like peptide-1 (GLP-1), is normally released by the intestine in response to the presence of food. This hormone acts like a messenger between the intestine and the pancreas to raise insulin levels, and therefore, lower blood sugars. Sitagliptin is effective in people with diabetes, however, this study is being done to determine if Sitagliptin is effective in people with high fasting glucose who do not yet have diabetes.

DETAILED DESCRIPTION:
Impaired fasting glucose (IFG) confers a high risk of progression to diabetes. Its pathogenesis has been an area of active investigation, with defects in insulin and glucagon secretion as well as insulin action likely to play a role. Several studies have suggested that the prediabetic and diabetic state are associated with alterations in circulating incretin concentrations. More recently, a large study of non-diabetic individuals demonstrated decreased GLP-1 concentrations after a glucose challenge in individuals with prediabetes but concluded that defects in GLP-1 secretion were unrelated to insulin secretion. In impaired glucose tolerance (IGT), defects in incretin-induced insulin secretion coexist with defects in glucose induced insulin secretion.

Worsening degrees of glucose tolerance are associated with decreased insulin secretion for the prevailing insulin action. Moreover early glucagon suppression is impaired in IGT. Since GLP-1 is an insulin secretagogue and suppresses glucagon, it is conceivable that defects in GLP-1 secretion could contribute to the pathogenesis of pre-diabetes. Inhibition of Dipeptidyl Peptidase-4 (DPP-4), an enzyme which rapidly degrades the incretin hormones, has been shown to be a useful therapeutic strategy in type 2 diabetes. DPP-4 inhibitors increase (model-calculated) insulin secretion and decrease glucagon concentrations resulting in a lowering of fasting (and postprandial) glucose concentrations in people with type 2 diabetes. Their effects in people with IFG are less certain. However, DPP-4 inhibitors provide an opportunity to directly examine the contribution of abnormal incretin concentrations to the pathogenesis of IFG, by raising concentrations of endogenous incretin hormones.

The current experiments tested this hypothesis by measuring insulin secretion and action and fasting and postprandial glucose turnover before and after 8 weeks of therapy with a DPP-4 inhibitor.

ELIGIBILITY:
Twenty four participants aged 35 to 70 years with impaired fasting glucose (100mg/dl-125 mg/dl) will be studied.

Inclusion Criteria:

* Males and females between the ages of 35-70.
* Good health as determined by past medical history,physical examination, vital signs, electrocardiogram and laboratory tests at the time of screening.
* Patients on diuretics or thyroid hormone therapy must be on a stable dose (at least 3 months prior to screening) and the maintenance dose may not be adjusted during the study.

Exclusion Criteria:

* Individuals with a body mass index less than 19 or greater than 40 kg/m^2, or a total weight > 130 kg, will be excluded from study.
* Subjects less than 35 years will not be studied in order to minimize the possibility of studying subjects with type 1 diabetes.
* No history of a) significant nephropathy, (i.e., plasma creatinine > 1.4 mg/dl in women and 1.5 mg/dl in men, and/or proteinuria); b) clinically significant atherosclerotic vascular disease (e.g., history of heart attack or angina); c) a known systemic illness.
* Pregnant or lactating females.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Bock G, Dalla Man C, Micheletto F, Basu R, Giesler PD, Laugen J, Deacon CF, Holst JJ, Toffolo G, Cobelli C, Rizza RA, Vella A. The effect of DPP-4 inhibition with sitagliptin on incretin secretion and on fasting and postprandial glucose turnover in subjects with impaired fasting glucose. Clin Endocrinol (Oxf). 2010 Aug;73(2):189-96. doi: 10.1111/j.1365-2265.2009.03764.x. Epub 2009 Dec 18. PMID 20039889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Impaired Fasting Glucose (IFG) not on treatment with glucose-lowering medication
Groups:
- Sitagliptin: People with impaired fasting glucose treated with sitagliptin 100mg once daily.
- Placebo: People with impaired fasting glucose treated with placebo once daily.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (2.5) | 54.1 (2.4) | 54.7 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Lowering of Fasting Glucose
Description: fasting glucose taken as the mean of blood glucose measured at -30, -20, -10 and 0 minutes prior to each inpatient meal study
Time Frame: 8 weeks
Population: Analysis was per protocol - all participants completed the intervention
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 11 | 11
mmol/l | 5.78 (0.12) | 5.83 (0.12)
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Paired comparisons (within groups) to examine differences between the baseline study and after 8-weeks of treatment were made using Student's two-tailed t-test for paired samples. Between-group comparisons were made using Student's two-tailed t-test for unpaired samples. Given the previously observed variation in fasting glucose; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Twelve weeks
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=11) | Placebo (N=11)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No